CLINICAL TRIAL: NCT00059748
Title: Studies of Natural History, Pathogenesis, and Outcomes in Autoimmune and Inflammatory Diseases Including Juvenile Dermatomyositis
Brief Title: Studies of the Natural History, Pathogenesis, and Outcome of Autoinflammatory Diseases Including Juvenile Dermatomyositis
Status: Recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030173; 03-AR-0173
Record Dates: First submitted 2003-05-05; First posted 2003-05-06 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-25

CONDITIONS: Autoinflammatory Disease; Juvenile Dermatomyositis
Keywords: Myositis; JDM; Immune Dysregulation; Skin Rash; Inflammation; Natural History
MeSH Terms: conditions — Dermatomyositis; Myositis; Exanthema; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected with autoinflammatory diseases: Subjects with known or suspected diagnosis of NOMID / CAPS, DIRA, CANDLE, SAVI, CRMO, Still s disease, Behcet s disease, JDM, and other autoinflammatory diseases.

SUMMARY:
Purpose:

The purpose of this protocol is 1. To comprehensively evaluate patients with autoinflammatory diseases clinically, genetically and immunologically at the autoinflammatory disease clinic at the NIH. 2. To follow patients with autoinflammatory Diseases that are genetically defined including Neonatal-Onset Multisystem Inflammatory Disease (NOMID), the most severe clinical phenotype of Cryopyrin-Associated Periodic Syndromes (CAPS), Deficiency of IL-1 Receptor Antagonist (DIRA), Chronic Atypical Neutrophilic Dermatosis with Lipodystrophy and Elevated temperatures (CANDLE), and STING-Associated Vasculopathy with onset in Infancy (SAVI), and those with genetically undefined autoinflammatory disorders to determine long-term disease outcomes. 3. To develop biomarkers that help us assess disease activity and response to treatment. 4. To assess the eligibility of affected patients for inclusion in ongoing and planned treatment protocols.

Goal: The goals of our studies are to understand the underlying immune dysregulation, to identify the genetic cause and to translate our findings into novel treatments that improve patients disease outcome.

Eligibility:

* Patients with known NOMID/CAPS, DIRA, CANDLE, SAVI, CRMO, Still's Disease, and with other yet undifferentiated autoinflammatory diseases.
* Healthy adult and pediatric relatives.
* Volunteers

Design:

Participants will be evaluated at the NIH for 2-5 days. All participants will have a detailed medical history, physical exam, blood tests and other evaluations depending on the extend of their autoinflammatory disease.

Participants may also expect the following assessments:

1. Clinical test that help assess organ damage and functional impact such as hearing vision, memory and learning tests.
2. Imaging studies to characterize the organ involvement of the inflammatory disease including: X-rays, CT scans, special MRIs, bone scans.
3. Laboratory evaluations including clinical markers of disease activity, research samples for genetic studies, and blood samples for cytokine/biomarker assessment, and gene expression profiling.<TAB>
4. Completion of questionnaires to assess disease activity and quality of life.
5. If indicated, other procedures may be administered that include: a lumbar puncture if CNS inflammation is suspected and a skin biopsy if skin inflammation is present. other gastrointestinal procedures as they are clinically indicated.
6. Patients my have a research skin biopsy taken.

Participants may return for a single follow-up visits or for long term-follow up depending on their disease and willingness to be followed long-term.

DETAILED DESCRIPTION:
Autoinflammatory multisystem diseases are a group of diseases that are characterized by recurrent episodes of systemic inflammation as well as organ specific inflammation that can involve the skin, eyes, joints, bones, serosal surfaces, inner ear, and brain. We study rare diseases including CANDLE (chronic atypical neutrophilic dermatosis with lipodystrophy and elevated temperatures) caused by mutations in proteasome components, and recently SAVI (STING associated vasculopathy with onset in infancy) caused by mutations in TMEM173, and juvenile dermatomyositis (JDM), which shares some phenotypic features as well as an interferon (IFN) signature with SAVI and CANDLE. Many additional autoinflammatory phenotypes have no genetic causes, including autoinflammatory disorders that are not even clinically defined. In this research protocol we seek to comprehensively evaluate affected patients clinically, genetically, immunologically, and endocrinologically. In addition we intend to evaluate long- term outcomes and biomarkers over the time of observations. Eligibility for ongoing and planned treatment protocols will be determined by screening patients in this protocol. We plan to evaluate patients on a consultative basis for other autoinflammatory diseases for possible enrollment into this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with CANDLE, SAVI, and JDM who are mutation positive for the disease or fulfill clinical criteria of the disease.
* Patients who fulfill criteria for definite or probable JDM
* Patients with other suspected autoinflammatory diseases
* There is:

  * 2 years old or older
  * Patients or their legal guardians need to be able and willing to give informed consent and a pediatric patient needs to be willing to assent to the protocol whenever possible.

Relatives of patients with autoinflammatory diseases or healthy volunteers may be included for genetic testing. The genetic evaluations will be conducted in collaboration with Dr. Fleisher's laboratory at the Clinical Center laboratory and other groups. We may also collect blood for serum and RNA analyses to establish a cohort of healthy controls that is matched in age, gender and ethnicity to the study patients. Skin biopsies for research may be requested from patients, patient relatives and healthy volunteers

EXCLUSION CRITERIA:

* Active malignancy or any medical condition that in the opinion of the investigator would warrant exclusion
* Inability to return for follow up visits
* Pregnancy
* Adults without the capacity to consent

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with auto inflammatory diseases
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2003-05-09 (Actual)

PRIMARY OUTCOMES:
Identification of disease pathogenesis | each visit
  Clinical, immunological, genetic and endocrinological characteristics of the disease

SECONDARY OUTCOMES:
To develop long term clinical and laboratory outcome parameters of multiorgan involvement in patients and evaluation of blood, body fluid, and tissue biomarkers during disease flares and quiescence. | each visit
  Subject is determined to be eligible or not eligible for enrollment onto a treatment or intervention protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Kim, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Rodriguez-Smith J, Lin YC, Tsai WL, Kim H, Montealegre-Sanchez G, Chapelle D, Huang Y, Sibley CH, Gadina M, Wesley R, Bielekova B, Goldbach-Mansky R. Cerebrospinal Fluid Cytokines Correlate With Aseptic Meningitis and Blood-Brain Barrier Function in Neonatal-Onset Multisystem Inflammatory Disease: Central Nervous System Biomarkers in Neonatal-Onset Multisystem Inflammatory Disease Correlate With Central Nervous System Inflammation. Arthritis Rheumatol. 2017 Jun;69(6):1325-1336. doi: 10.1002/art.40055. Epub 2017 May 10. PMID 28118536
- [Derived] Chang Z, Spong CY, Jesus AA, Davis MA, Plass N, Stone DL, Chapelle D, Hoffmann P, Kastner DL, Barron K, Goldbach-Mansky RT, Stratton P. Anakinra use during pregnancy in patients with cryopyrin-associated periodic syndromes (CAPS). Arthritis Rheumatol. 2014 Nov;66(11):3227-32. doi: 10.1002/art.38811. PMID 25223501
- [Derived] Liu Y, Jesus AA, Marrero B, Yang D, Ramsey SE, Sanchez GAM, Tenbrock K, Wittkowski H, Jones OY, Kuehn HS, Lee CR, DiMattia MA, Cowen EW, Gonzalez B, Palmer I, DiGiovanna JJ, Biancotto A, Kim H, Tsai WL, Trier AM, Huang Y, Stone DL, Hill S, Kim HJ, St Hilaire C, Gurprasad S, Plass N, Chapelle D, Horkayne-Szakaly I, Foell D, Barysenka A, Candotti F, Holland SM, Hughes JD, Mehmet H, Issekutz AC, Raffeld M, McElwee J, Fontana JR, Minniti CP, Moir S, Kastner DL, Gadina M, Steven AC, Wingfield PT, Brooks SR, Rosenzweig SD, Fleisher TA, Deng Z, Boehm M, Paller AS, Goldbach-Mansky R. Activated STING in a vascular and pulmonary syndrome. N Engl J Med. 2014 Aug 7;371(6):507-518. doi: 10.1056/NEJMoa1312625. Epub 2014 Jul 16. PMID 25029335
- [Derived] Aksentijevich I, Masters SL, Ferguson PJ, Dancey P, Frenkel J, van Royen-Kerkhoff A, Laxer R, Tedgard U, Cowen EW, Pham TH, Booty M, Estes JD, Sandler NG, Plass N, Stone DL, Turner ML, Hill S, Butman JA, Schneider R, Babyn P, El-Shanti HI, Pope E, Barron K, Bing X, Laurence A, Lee CC, Chapelle D, Clarke GI, Ohson K, Nicholson M, Gadina M, Yang B, Korman BD, Gregersen PK, van Hagen PM, Hak AE, Huizing M, Rahman P, Douek DC, Remmers EF, Kastner DL, Goldbach-Mansky R. An autoinflammatory disease with deficiency of the interleukin-1-receptor antagonist. N Engl J Med. 2009 Jun 4;360(23):2426-37. doi: 10.1056/NEJMoa0807865. PMID 19494218
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-AR-0173.html